CLINICAL TRIAL: NCT05111080
Title: Partial PTEN Deletion and Its Relation to Clinicopathological Characteristics in Breast Cancer Patients
Brief Title: Partial PTEN Deletion in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: principle investigator (Unknown)
Responsible Party: Principal Investigator, Fatma Refaat Ibrahim Ismail, resident doctor, Assiut University
Other Study IDs: FISH in breast cancer
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: PTEN Gene Deletion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Detection of chromosome 10q23 deletion including PTEN locus in breast cancer patients.
* Correlation between PTEN deletion and clinicopathological characteristics in breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common carcinoma detected in women, accounting for about one fifth of new cancer cases in females. In Egypt breast cancer is the most common malignancy in women, accounting for 38,8% of cancers in this population, with the estimated number of breast cancer cases nearly 22700 in 2020 and forecasted to be approximately 46000 in 2050. Surgical removal of the cancer represents the standard of care followed by radiation and adjuvant therapy in patients considered to be at particular risk for systemic disease. Estimation of prognosis is of vital importance for tailoring adjuvant therapy in individual breast cancer patients. Conventional pathological parameters such as histological grade, tumor size and presence of lymph node metastasis are not accurate enough to select subsets of patients who are at sufficiently low risk of progression to be spared extensive adjuvant therapy without compromising the prognosis. Much hope is placed on cytogenetic features analysis which might help to improve prediction of patient prognosis.

Fluorescence in situ hybridization (FISH) is a molecular cytogenetic technique that enables the detection of genetic abnormalities such as gene amplification, deletions, and chromosomal rearrangements.

Deletions of chromosome 10q23 including the PTEN (phosphatase and tensin homolog) locus are known to occur in breast cancer patients. The PTEN gene is a phosphatase which metabolises PIP3, the lipid product of PI 3-kinase, directly opposing the activation of the oncogenic PI3K/AKT/mTOR signalling network. Inactivation of PTEN leads to constitutively activated levels of AKT, thus promoting cell growth, proliferation, survival and migration through multiple downstream effectors. PTEN is one of the most frequently deleted genes in various human cancer types. In breast cancer, the frequency of PTEN deletions or reduced expression varies from 4 % to 63 %.

ELIGIBILITY:
Inclusion Criteria:

* all stages of breast cancer in females.

Exclusion Criteria:

* breast cancer in males.

Min Age: 20 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All stages of female patients with breast cancer. Median age was 63 (range 20-100) years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Detection of chromosome 10q23 deletion including PTEN locus in breast cancer patients. | baseline
  Correlation between PTEN deletion and clinicopathological characteristics in breast cancer patients.

REFERENCES:
- [Background] Young PA, Kaiser II. Aminoacylation of Escherichia coli cysteine tRNA by selenocysteine. Arch Biochem Biophys. 1975 Dec;171(2):483-9. doi: 10.1016/0003-9861(75)90057-0. No abstract available. PMID 963